CLINICAL TRIAL: NCT01182571
Title: Exploration of Fatigue ,Uncertainty ,Depression and Quality of Life in Heart Transplantation Recipients
Brief Title: Exploration of Fatigue, Uncertainty, Depression and Quality of Life in Heart Transplantation Recipients
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Shun,Shiow-Ching, Department of Nursing, College of Medicine, National Taiwan University
Other Study IDs: 200808050R
Record Dates: First submitted 2009-08-24; First posted 2010-08-17 (Estimated); Last update posted 2010-08-30 (Estimated); Status verified 2010-08

CONDITIONS: Heart Transplantation
Keywords: Heart Transplantation; Symptom Distress; Fatigue; Depression; Quality Of Life.
MeSH Terms: conditions — Fatigue; Depression

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- heart transplantation

SUMMARY:
The purpose of this study is to explore the fatigue, uncertainty, depression and quality of life in heart transplant recipients, and associated factors of quality of life .

DETAILED DESCRIPTION:
The purpose of this study is to explore the symptom distress, fatigue, depression, uncertainty, and quality of life in heart transplant recipients, and associated factors of quality of life (QOL). The eligible patients are (1)who undergone heart transplantation were recruited from the Department of Cardiac Surgery, Nation Taiwan University Hospital,(2)18 year old or older. A set of questionnaire with the Transplant Symptom Frequency and Symptom Distress Scale, Hospital Anxiety and Depression Scale (HADS) , Fatigue Symptom Inventory (FSI), Mishel's Uncertainty Scale, and 12-item Short-Form Health Survey (SF-12) were used to collected symptom distress, fatigue, depression, uncertainty, and QOL .

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of heart transplantation
* Adults 18 years of age

Exclusion Criteria:

* The woman who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The outpatients who undergone heart transplantation were recruited from the Department of Cardiac Surgery
Sampling Method: Non-Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2008-10; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
The SF12 Health survey | 1 month
  It was used to measure quality of life
Transplant Symptom Frequency and Symptom Distress Scale | 1 week
  it was used to measure symptom distress.
Fatigue Symptom Inventory | 1 week
  It was used to measure level of fatigue.
Hospital Anxiety and Depression Scale (HADS) | 1month
  It was used to measure level of anxiety and depression.
Illness Uncertainty Scale | 1 month
  It was used to measure level of uncertainty.

CONTACTS AND LOCATIONS:
Overall Officials: Shiow-Ching Shun, PhD, Principal Investigator — National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan